CLINICAL TRIAL: NCT00315744
Title: Steroid-sparing Management of the Salmeterol/Fluticasone 50/100µg b.i.d. Combination Compared to Fluticasone 200µg b.i.d. in Children and Adolescents With Moderate Asthma
Brief Title: Viapaed Study In Children And Adolescents With Asthma
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: 102318
Record Dates: First submitted 2006-04-17; First posted 2006-04-19 (Estimated); Last update posted 2017-10-19 (Actual); Status verified 2017-10

CONDITIONS: Asthma
Keywords: moderate asthma; fluticasone; children; salmeterol; steroid-sparing; Asthma
MeSH Terms: conditions — Asthma | interventions — Fluticasone-Salmeterol Drug Combination; Fluticasone; Salmeterol Xinafoate; Albuterol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Subjects receiving salmeterol/fluticasone (Experimental): Eligible subjects will receive 60 individual doses of the salmeterol 50 microgram/ fluticasone 100 microgram combination. Subjects will also receive placebo.
  Interventions: Drug: Salmeterol/fluticasone; Drug: Salbutamol
- Subjects receiving fluticasone (Active Comparator): Eligible subjects will receive 60 individual fluticasone 100 microgram doses each.
  Interventions: Drug: Fluticasone propionate; Drug: Salbutamol

INTERVENTIONS:
Drug: Salmeterol/fluticasone — Salmeterol/ fluticasone are a type of long acting beta-agonist (LABA). Salmeterol 50 microgram/ fluticasone 100 microgram combination will be administered to eligible subjects via inhalation route.
  Arms: Subjects receiving salmeterol/fluticasone
Drug: Fluticasone propionate — Fluticasone propionate is a type of LABA. Fluticasone 100 microgram dose will be administered to eligible subjects via inhalation route.
  Other Names: Salmeterol; SERETIDE
  Arms: Subjects receiving fluticasone
Drug: Salbutamol — Salbutamol metered dose inhaler will be provided to all subjects as a rescue medication.

SUMMARY:
Asthmatic children who remain symptomatic on inhaled corticosteroids (ICS) require an adjustment of their asthma therapy. Current guidelines suggest that the treatment options are either an increased dose of inhaled corticosteroid or the addition of other therapy such as a long-acting beta-agonist (LABA). In the pediatric age range, major concerns with respect to high dose ICS therapy are growth retardation and the suppression of the hypothalamic-pituitary-adrenocortical (HPA) axis. Previous studies in adults have shown that a combination product that included a LABA as well as the ICS allowed to reduce the steroid dose and was still at least as effective in achieving asthma control as treatment with a higher dose of ICS. These treatment options shall be compared in the present study. Children who remain symptomatic while inhaling 100 µg fluticasone (FP) twice daily shall be randomized to receive the salmeterol/ fluticasone combination product, Viani (SERETIDE) 50/100 µg, or fluticasone 200 µg as a comparator drug, inhaled twice daily via the DISKUS for a period of eight weeks.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 4 to 16 years with an established history of perennial asthma.
* Subjects who are treated with an inhaled corticosteroid according to BDP (budesonide) 200-400 µg/day or equivalent during the last 4 weeks before run-in.
* 15 minutes after inhaling 200µg of salbutamol, reversible increase in FEV1 of at least 12% of the pre-dose value.
* Willingness to substitute previous controller medication on the twice daily inhalation of fluticasone 100µg bid via DISKUS®.
* Subjects/guardians who have given written informed consent to participate in the study.
* Subjects /guardians who are able to understand and complete a diary record card (DRC).
* Subjects who are able to use a Mini-Wright Peak Flow meter.
* Sexually active female adolescents must use adequate contraception.
* Willingness to refrain from any other controller medication (including anti-leukotrienes) or from regular use of short-acting beta agonists or anticholinergics during the treatment period.

Ages: 4 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 285 (Actual)
Dates: Start 2004-11-04 (Actual); Primary Completion 2007-04-12 (Actual); Study Completion 2007-04-12 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in mean morning peak expiratory flow (PEF) | Baseline up to Week 8
  The PEF is a person's maximum speed of expiration. PEF will be measured using a mini wright peak flow meter and will be documented daily at morning in the diary of subjects

SECONDARY OUTCOMES:
Daily Asthma symptom score | Up to Week 8
  Asthma symptoms will be recorded separately for night and day using 2 symptom scores. Symptoms included will be coughing, wheezing, shortness of breath, feeling of tightness in the chest and nocturnal waking due to 1 or more of these symptoms. Score will range from 0-4 where 0 = no complaints and 4= person could not sleep due to asthma symptoms.
Number of calendar days without asthma symptoms | Up to Week 8
  Number of calendar days without asthma symptoms will be defined as the sum of all days for which the patient documented an asthma symptom score of 0 (no complaints) for the day and the previous night.
Number of necessary administrations of salbutamol | Up to Week 8
  The number of necessary administrations of salbutamol will be documented daily by subjects in the diary.
Number of weeks with good asthma control | Up to Week 8
  One week of well controlled asthma will be defined by fulfilling the following criteria: at least 2 of the following criteria (type A): symptoms with a symptom score >1 on at most 2 days, use of rescue medication maximally 4 x per week, morning PEF daily >=80% of the predicted normal value and all the following criteria (type B): no nocturnal waking due to bronchial asthma, no exacerbations, no out-patient or hospitalized emergency treatment due to asthma, no adverse events due to administration of the study medication which would have necessitated a change of treatment, no intolerance or refusal of study medication
Change in forced vital capacity (FVC) in % of reference value | Up to Week 8
  FVC is the amount of air which can be forcibly exhaled from the lungs after taking the deep breath.
Change in forced expiratory volume in 1 second (FEV1) in % of reference value | Up to Week 8
  FEV1 is the volume of air exhaled under forced conditions in 1 second.
Change in peak expiratory flow rate (PEFR) in % of reference value | Up to Week 8
  PEFR is a person's maximum speed of expiration.
Change in mean morning peak flow in % of reference value | Up to Week 8
  The PEF is a person's maximum speed of expiration. PEF will be measured using a mini wright peak flow meter
Percentage of subjects with a peak flow variability of 20% | Up to Week 8
  Morning versus evening peak flow will be calculated and compared.
Number of subject withdrawals due to asthma exacerbations | Up to Week 8
  Asthma exacerbations are acute or sub acute episodes, which are characterized by a progressive increase in one or more typical asthma symptoms.
Number of subjects with adverse events (AEs) | Up to Week 8
  An AE is any untoward medical occurrence in a clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (75):
- Germany (75):
  - GSK Investigational Site, Bad Krozingen, Baden-Wurttemberg
  - GSK Investigational Site, Bönnigheim, Baden-Wurttemberg
  - GSK Investigational Site, Ettenheim, Baden-Wurttemberg
  - GSK Investigational Site, Heidelberg, Baden-Wurttemberg
  - GSK Investigational Site, Kehl, Baden-Wurttemberg
  - GSK Investigational Site, Konstanz, Baden-Wurttemberg
  - GSK Investigational Site, Mannheim, Baden-Wurttemberg
  - GSK Investigational Site, Pfullendorf, Baden-Wurttemberg
  - GSK Investigational Site, Schwäbisch Hall, Baden-Wurttemberg
  - GSK Investigational Site, Schwetzingen, Baden-Wurttemberg
  - GSK Investigational Site, Sinsheim, Baden-Wurttemberg
  - GSK Investigational Site, Stuttgart, Baden-Wurttemberg
  - GSK Investigational Site, Tauberbischofsheim, Baden-Wurttemberg
  - GSK Investigational Site, Tuttlingen, Baden-Wurttemberg
  - GSK Investigational Site, Villingen-Schwenningen, Baden-Wurttemberg
  - GSK Investigational Site, Welzheim, Baden-Wurttemberg
  - GSK Investigational Site, Bobingen, Bavaria
  - GSK Investigational Site, Forchheim, Bavaria
  - GSK Investigational Site, Freising, Bavaria
  - GSK Investigational Site, Kaufbeuren, Bavaria
  - GSK Investigational Site, Lauf, Bavaria
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Nördlingen, Bavaria
  - GSK Investigational Site, Nuremberg, Bavaria
  - GSK Investigational Site, Olching, Bavaria
  - GSK Investigational Site, Pegnitz, Bavaria
  - GSK Investigational Site, Rosenheim, Bavaria
  - GSK Investigational Site, Frankfurt (Oder), Brandenburg
  - GSK Investigational Site, Schwedt, Brandenburg
  - GSK Investigational Site, Braunfels, Hesse
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Kassel, Hesse
  - GSK Investigational Site, Niedernhausen, Hesse
  - GSK Investigational Site, Wetzlar, Hesse
  - GSK Investigational Site, Wiesbaden, Hesse
  - GSK Investigational Site, Belm, Lower Saxony
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Lüneburg, Lower Saxony
  - GSK Investigational Site, Osnabrück, Lower Saxony
  - GSK Investigational Site, Aachen, North Rhine-Westphalia
  - GSK Investigational Site, Bielefeld, North Rhine-Westphalia
  - GSK Investigational Site, Bochum, North Rhine-Westphalia
  - GSK Investigational Site, Bottrop, North Rhine-Westphalia
  - GSK Investigational Site, Detmold, North Rhine-Westphalia
  - GSK Investigational Site, Dortmund, North Rhine-Westphalia
  - GSK Investigational Site, Duisburg, North Rhine-Westphalia
  - GSK Investigational Site, Düsseldorf, North Rhine-Westphalia
  - GSK Investigational Site, Essen, North Rhine-Westphalia
  - GSK Investigational Site, Euskirchen, North Rhine-Westphalia
  - GSK Investigational Site, Gütersloh, North Rhine-Westphalia
  - GSK Investigational Site, Halle, North Rhine-Westphalia
  - GSK Investigational Site, Kempen, North Rhine-Westphalia
  - GSK Investigational Site, Kleve-Materborn, North Rhine-Westphalia
  - GSK Investigational Site, Krefeld, North Rhine-Westphalia
  - GSK Investigational Site, Minden, North Rhine-Westphalia
  - GSK Investigational Site, Neuss, North Rhine-Westphalia
  - GSK Investigational Site, Oberhausen, North Rhine-Westphalia
  - GSK Investigational Site, Remscheid, North Rhine-Westphalia
  - GSK Investigational Site, Wesel, North Rhine-Westphalia
  - GSK Investigational Site, Willich, North Rhine-Westphalia
  - GSK Investigational Site, Koblenz, Rhineland-Palatinate
  - GSK Investigational Site, Mainz, Rhineland-Palatinate
  - GSK Investigational Site, Trier, Rhineland-Palatinate
  - GSK Investigational Site, Cossebaude, Saxony
  - GSK Investigational Site, Döbeln, Saxony
  - GSK Investigational Site, Dresden, Saxony
  - GSK Investigational Site, Leipzig, Saxony
  - GSK Investigational Site, Wurzen, Saxony
  - GSK Investigational Site, Flensburg, Schleswig-Holstein
  - GSK Investigational Site, Geesthacht, Schleswig-Holstein
  - GSK Investigational Site, Harrislee, Schleswig-Holstein
  - GSK Investigational Site, Friedrichsfelde, State of Berlin
  - GSK Investigational Site, Neuhaus am Rennweg, Thuringia
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Hamburg

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Gappa M, Zachgo W, von Berg A, Kamin W, Stern-Strater C, Steinkamp G; VIAPAED Study Group. Add-on salmeterol compared to double dose fluticasone in pediatric asthma: a double-blind, randomized trial (VIAPAED). Pediatr Pulmonol. 2009 Nov;44(11):1132-42. doi: 10.1002/ppul.21120. PMID 19824054
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: 102318 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 102318 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 102318 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 102318 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 102318 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 102318 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register